CLINICAL TRIAL: NCT03839316
Title: The Effect of Bihemispheric Transcranial Direct Current Stimulation Therapy on Upper Extremity Motor Functions in Stroke Patients
Brief Title: Effects of Bihemispheric Transcranial Direct Current Stimulation on Motor Function in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Dilek Cetinkaya Alisar, physical and rehabilitation medicine trainee, Baskent University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KA15/271
Record Dates: First submitted 2019-02-11; First posted 2019-02-15 (Actual); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Stroke; Upper Extremity Paresis; Transcranial Direct Current Stimulation
Keywords: Cortical stimulation; Motor function; Rehabilitation; Stroke
MeSH Terms: conditions — Stroke; Paresis | interventions — Transcranial Direct Current Stimulation; Occupational Therapy

STUDY DESIGN:
Intervention Model Description: The aim of the study is to evaluate and compare the effect of tDCS plus conventional physiotherapy and occupational therapy to sham tDCS plus conventional physiotherapy and occupational therapy on upper extremity motor function in patients with subacute stroke was aimed in our study.
  32 patients will be randomly assigned to one of two groups in parallel for the duration of the study: bihemispheric tDCS (n:16), or sham tDCS (n:16). In addition to a conventional physiotherapy and occupational therapy program, bihemispheric tDCS application will be applied to one group and sham tDCS applied to the second group. A constant current stimulator(ZMI Electronics Limited,Taiwan,2012) will be used for the application of tDCS. In both groups, the tDCS application will be started simultaneously with the occupational therapy session and will last for thirty minutes.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tDCS group (Active Comparator): Sixteen stroke patient receiving bihemispheric tDCS in addition to a conventional physiotherapy (PT) and occupational therapy (OT) program for five consecutive days per week for a three week period (a total of fifteen sessions).
  The one hour long conventional PT sessions will include an upper extremity range of motion, strengthening and neurofacilitation exercise program. The one hour long OT sessions will include task specific exercises chosen according to the patient's functional status, including activities aimed at improving gross and fine motor function of the upper extremities.
  The tDCS application will be applied at the beginning of each OT session and will be continued for a total of thirty minutes at 2 mA.
  Interventions: Device: tDCS
- Sham group (Sham Comparator): Sixteen stroke patient receiving a conventional PT and OT program and sham tDCS for 5 consecutive days per week for a 3 week period ( a total of 15 sessions). The one hour long conventional PT and OT sessions will be the same as in the tDCS group. For sham tDCS, electrode application and positioning will be the same as the intervention group and will be applied at the beginning of each OT session as previously described. The current will initially be increased up to 2 mA, so to provide the typical initial tingling sensation, and slowly decreased over 30 seconds and consequently switched off. The electrodes will be removed after a total of thirty minutes.
  Interventions: Device: sham tDCS

INTERVENTIONS:
Device: tDCS — A constant current stimulator (ZMI Electronics LTD.,Taiwan,2012) will be used through 2 saline-soaked surface gel-sponge electrodes (22 cm2 active area). Real stimulation consisting of thirty minutes of 2 mA direct current with the anode placed over the ipsilesional and the cathode over the contralesional motor cortex (C3 and C4 of the international 10-20 EEG electrode system).
  Other Names: Conventional physiotherapy and occupational therapy
  Arms: tDCS group
Device: sham tDCS — For sham tDCS, the same electrode positions were used. The current was ramped up to 2 mA and slowly decreased over 30 seconds to ensure the typical initial tingling sensation
  Other Names: Conventional physiotherapy and occupational therapy
  Arms: Sham group

SUMMARY:
Motor impairment (impairment of movement) due to stroke is one of the leading disabilities in adults. In addition to established means of facilitating motor recovery after stroke such as physical and occupational therapy, a variety of experimental rehabilitation approaches have been tested. Although there have been significant advances in stroke rehabilitation with these techniques and treatments, research on this subject is continuing. Recent studies have focused on non-invasive brain stimulation techniques. Transcranial magnetic stimulation (TMS) or transcranial direct current stimulation (tDCS) therapies, which are methods of non-invasive brain stimulation that may be effective on cerebral remodelling, aim to reestablish the disturbed balance between the anatomic areas of the brain seen in stroke patients.

The primary aim of this study is to evaluate the effectiveness of bihemispheric transcranial direct current stimulation (tDCS) applications on the upper extremity motor functions of patients with stroke.

DETAILED DESCRIPTION:
Motor impairment due to ischemic and hemorrhagic stroke is one of the leading disabilities in adults. In addition to established means of facilitating motor recovery after stroke such as physical and occupational therapy, a variety of experimental rehabilitation approaches have been tested. Recent developments include noninvasive brain stimulation techniques such as repetitive transcranial magnetic stimulation (rTMS) and transcranial direct current stimulation (tDCS). The use of these tools is based on neurophysiologic studies demonstrating an imbalance of interhemispheric interactions which appears to interfere with the recovery process.

The model of interhemispheric imbalance provides a framework for developing hypotheses based on its 2 facets: 1) upregulating excitability of intact portions of the ipsilesional motor cortex and 2) downregulating excitability of the contralesional motor cortex to modulate its unrestrained inhibitory influence on ipsilesional regions. Studies to date have shown have shown the beneficial effects of tDCS on motor skills and motor learning.

Bihemispheric tDCS may potentiate the effects of anodal stimulation to the lesional hemisphere through additional modulation of interhemispheric interactions via cathodal stimulation to the contralesional motor cortex.

The primary aim of this prospective, randomized, sham controlled study is to evaluate the effectiveness of bihemispheric transcranial direct current stimulation (tDCS) applications on the upper extremity motor functions of patients with stroke.

ELIGIBILITY:
Inclusion Criteria:

1. 18-75 years old, female or male
2. Clinical evaluation consistent with hemiplegia
3. First time stroke with brain computerized tomography (CT) and / or magnetic resonance imaging (MRI) findings consistent with stroke
4. At least 3 months since stroke onset
5. Presence of a stable medical condition
6. Preserved cognitive function as determined by a mini mental state examination score of 23 and above

Exclusion Criteria:

1. Presence of a sensory aphasia
2. Presence of neglect syndrome
3. A history of epilepsy
4. Presence of a pacemaker
5. Previous history of stroke
6. History of previous cranial surgery
7. Presence of a brain tumour
8. Presence of an intracranial metallic implant
9. Marked hearing / visual impairment
10. Presence of severe spasticity (grade 3-4 according to the modified Ashworth scale)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Change in upper extremity impairment | Before treatment sessions begin and 1 week after fifteen treatment sessions have been completed (three weeks after the initial onset of treatment).
  The Fugl-Meyer Upper Extremity (FMUE) Scale is a widely used and highly recommended stroke-specific, performance-based measure of impairment. It is designed to assess reflex activity, movement control and muscle strength in the upper extremity of people with post-stroke hemiplegia. It has been extensively used as an outcome measure in rehabilitation trials and to record poststroke recovery, particularly in the USA.
  The FMUE Scale comprises 33 items, each scored on a scale of 0 to 2, where 0 = cannot perform, 1 = performs partially and 2 = performs fully. It is free, requires only household items for testing, and takes up to 30 minutes to administer.The total score ranges from 0-66 where 66. The higher the score the less the level of impairment.

SECONDARY OUTCOMES:
Change in functionality | Before treatment sessions begins and 1 week after fifteen treatment sessions have been completed (three weeks after the initial onset of treatment)
  The Functional Independence Measure (FIM) is an 18-item seven level ordinal scale of physical, psychological and social function.The tool is used to assess a patient's level of functionality as well as change in patient status in response to rehabilitation or medical intervention. 13 of the 18 items of the FIM assess motor function and provide a 'motor score', the remaining five questions assess communication and social skills and provide a 'cognitive score' . Each item is scored from 1=complete dependence of task to 7=complete independence of task. The lowest possible attainable total score is 18 and the highest possible attainable total score is 126. The higher the score the higher the level of independence. When considering the subscores, the lowest possible attainable motor score is 13 and the highest is 91. The lowest possible attainable cognitive subscore is 5 and the highest is 35.
Change in motor activity | Before treatment sessions begins and 1 week after fifteen treatment sessions have been completed (three weeks after the initial onset of treatment)
  The Brunnstrom Stages of Stroke Recovery is a test that evaluates the motor development of stroke patients. In 1966, Signe Brunnstrom identified the stages of motor development observed in a large number of hemiplegic patients. In this staging, the hemiplegic upper extremity, lower extremity and hand are evaluated separately and the motor development of these three areas are staged from 1-6. The lowest stage according to this staging system is stage 1 (flask, no movement); the highest stage is stage 6 (normal motor function). Higher Brunnstrom stages indicate better motor development.

CONTACTS AND LOCATIONS:
Overall Officials: Seyhan Sozay, MD, Study Director — Baskent University Faculty of Medicine
Locations (1):
- Baskent University Faculty of Medicine,Ankara Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after identification (text, tables, figures and appendices) will be made available
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available for 6 months following article publication
Access Criteria: The data will be shared with researchers providing a methodologically sound proposal Proposals should be directed to drdilekalisar@gmail.com. To gain access, data requestors will need to sign a data access agreement. Data will be accessible for a period of one year.

REFERENCES:
- [Background] Lindenberg R, Renga V, Zhu LL, Nair D, Schlaug G. Bihemispheric brain stimulation facilitates motor recovery in chronic stroke patients. Neurology. 2010 Dec 14;75(24):2176-84. doi: 10.1212/WNL.0b013e318202013a. Epub 2010 Nov 10. PMID 21068427
- [Background] Tedesco Triccas L, Burridge JH, Hughes AM, Pickering RM, Desikan M, Rothwell JC, Verheyden G. Multiple sessions of transcranial direct current stimulation and upper extremity rehabilitation in stroke: A review and meta-analysis. Clin Neurophysiol. 2016 Jan;127(1):946-955. doi: 10.1016/j.clinph.2015.04.067. Epub 2015 May 4. PMID 25998205
- [Background] Elsner B, Kugler J, Mehrholz J. Transcranial direct current stimulation (tDCS) for upper limb rehabilitation after stroke: future directions. J Neuroeng Rehabil. 2018 Nov 15;15(1):106. doi: 10.1186/s12984-018-0459-7. PMID 30442158
- [Background] Chhatbar PY, Ramakrishnan V, Kautz S, George MS, Adams RJ, Feng W. Transcranial Direct Current Stimulation Post-Stroke Upper Extremity Motor Recovery Studies Exhibit a Dose-Response Relationship. Brain Stimul. 2016 Jan-Feb;9(1):16-26. doi: 10.1016/j.brs.2015.09.002. Epub 2015 Sep 7. PMID 26433609
- [Background] Fusco A, De Angelis D, Morone G, Maglione L, Paolucci T, Bragoni M, Venturiero V. The ABC of tDCS: Effects of Anodal, Bilateral and Cathodal Montages of Transcranial Direct Current Stimulation in Patients with Stroke-A Pilot Study. Stroke Res Treat. 2013;2013:837595. doi: 10.1155/2013/837595. Epub 2013 Jan 8. PMID 23365790
- [Background] Hall KM, Hamilton BB, Gordon WA, Zasler ND. Characteristics and comparisons of functional assessment indices: Disability rating scale, functional independence measure and functional assessment measure. Journal of Head Trauma Rehabilitation 8(2):60-74, 1993
- [Background] Sullivan KJ, Tilson JK, Cen SY, Rose DK, Hershberg J, Correa A, Gallichio J, McLeod M, Moore C, Wu SS, Duncan PW. Fugl-Meyer assessment of sensorimotor function after stroke: standardized training procedure for clinical practice and clinical trials. Stroke. 2011 Feb;42(2):427-32. doi: 10.1161/STROKEAHA.110.592766. Epub 2010 Dec 16. PMID 21164120